CLINICAL TRIAL: NCT03060330
Title: Obstructed Defecation Caused by Rectal Prolapse and Rectocele: Laparoscopic Ventral Rectopexy Alone Versus Laparoscopic Ventral Rectopexy Combined With Stapled Trans-anal Rectal Resection
Brief Title: Laparoscopic Ventral Mesh Rectopexy Combined With or Without Stapled Trans-anal Rectal Resection for Obstructed Defecation Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Tao Fu, Chief of Department of Gastrointestinal Surgery II, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LVMRSTARRODS2017
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Defecation Syndrome; Chronic Constipation; Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVMR (Experimental): Modified Laparoscopic Ventral Mesh Rectopexy
  Interventions: Procedure: Modified Laparoscopic Ventral Mesh Rectopexy
- LVMR with STARR (Experimental): Modified Laparoscopic Ventral Mesh Rectopexy Combined with Stapled Trans-anal Rectal Resection
  Interventions: Procedure: Modified Laparoscopic Ventral Mesh Rectopexy Combined with Stapled Trans-anal Rectal Resection

INTERVENTIONS:
Procedure: Modified Laparoscopic Ventral Mesh Rectopexy — This group will undergo modified laparoscopic ventral mesh rectopexy alone
  Arms: LVMR
Procedure: Modified Laparoscopic Ventral Mesh Rectopexy Combined with Stapled Trans-anal Rectal Resection — This group will undergo modified laparoscopic ventral mesh rectopexy combined with modified stapled trans-anal rectal resection
  Arms: LVMR with STARR

SUMMARY:
Obstructed defecation syndrome (ODS) is a common problem in women. Rectal prolapse and rectocoele are frequently identified in patients with ODS. Surgery is the only definite treatment for those patients and is preferably performed minimally invasive. The most used procedures are laparoscopic ventral mesh rectopexy (LVMR) and stapled trans-anal rectal resection (STARR). However, high-level prospective studies on treatment strategies for ODS currently are lacking and, thus, no consensus exist regarding the optimal treatment for patients with ODS. This study aimed to compare LVMR alone and LVMR combined with STARR evaluating functional and anatomical results.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by obstructed defecation with a minimum ODS score of 10
* External rectal prolapse or high-grade internal rectal prolapse
* Often experience excessive straining, sense of incomplete evacuation, and/or prolonged time for complete evacuation when attempting a bowel movement
* Have experienced ODS symptoms for at least 12 months prior to enrollment
* Failure of at least 6 months of medical therapy
* American Society of Anesthesiologists (ASA) score of no more than 3

Exclusion Criteria:

* Slow transit constipation
* Anismus resistant to conventional treatment
* No demonstrable pelvic anatomical problem
* Previous rectal or anal surgery
* Recto-vaginal fistula
* Pregnancy
* Previous pelvic radiotherapy
* Severe proctitis or significant rectal fibrosis
* Evidence of colorectal neoplasia, carcinoma, or inflammatory bowel disease
* Perineal infection
* High-grade endometriosis
* Morbid obesity
* A hostile abdomen
* Psychological instability

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in the ODS score (ODS-S) | Baseline and 12 months after surgery
  The primary outcome measure will be the change in total ODS score (ODS-S) measured at 12 months after surgery.

SECONDARY OUTCOMES:
Postoperative complications | 0 to 12 months after surgery
  Monitoring of complications started in the hospital and is followed up in the outpatient setting until 12 months after surgery.
Changes in the Patient Assessment of Constipation- Quality of Life score (PAC-QoL) | Baseline, 1, 3, 6, and 12 months after surgery
  This is a measure of efficacy.
Changes in Health-Related Quality of Life | Baseline, 1, 3, 6, and 12 months after surgery
  SF-36 version 1 will be used to measure changes in the health-related quality of life. This is a measure of efficacy.
Changes in Cleveland Clinic Fecal Incontinence Score (CCFI) | Baseline, 1, 3, 6, and 12 months after surgery
  This is a measure of efficacy.
Changes in Fecal Incontinence Quality of Life Scale (FIQoL) | Baseline, 1, 3, 6, and 12 months after surgery
  This is a measure of efficacy.
Radiological outcome as assessed by defecography | Baseline and 12 months after surgery
  This is a measure of efficacy.
Changes in the ODS score (ODS-S) | Baseline, 1, 3, 6, and 12 months after surgery
  This is a measure of efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery II, Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No